CLINICAL TRIAL: NCT00878176
Title: Sacral Neuromodulation Test With Bilateral First Stage Tined Lead Procedure in Patients With Non-obstructive Urinary Retention: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MEC 09-2-005
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2009-09

CONDITIONS: Urinary Retention
Keywords: sacral neuromodulation therapy; urinary retention; screening; non obstructive urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): (Crossover study)
  Interventions: Procedure: First stage tined lead procedure

INTERVENTIONS:
Procedure: First stage tined lead procedure — bilateral first stage tined lead placement

SUMMARY:
The objective of this study is to determine whether bilateral sacral nerve stimulation with First stage tined lead placement test is more effective than unilateral stimulation, among patients with non obstructive urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent
* Patients (male and female), aged between 18-70 years, with non obstructive urinary retention.

Two specific subcategories of retention are included

1. Incomplete voiding or incomplete retention (>100 cc residual) such as hesitancy or intermittency, that are due to an acontractile detrusor or due to urethral sphincter overactivity. The overactivity of the sphincter may occur in absence of detrusor contraction and may be the cause of the lack of detrusor activity.
2. Complete retention. These individuals are completely unable to void.

All patients must have the potential for storing an adequate volume of urine:

i.e., at least 100 ml

Exclusion Criteria:

* Known psychiatric disorders
* Current or plans of pregnancy
* Known neurologic diseases or impairment; including DM (severe or uncontrolled diabetes; or diabetes with peripheral nerve involvement), spinal cord injury, MS
* Reiter's syndrome
* Concomitant medical conditions that would limit the success of the procedure such as: active degenerative disc disease, spinal cord injury< 6 months old, bleeding complications, CVA< 6 months old etc.
* Extra urethral incontinence
* Pelvic pain of uncertain etiology that is not associated with a voiding dysfunction or where pelvic pain is the primary complaint/ diagnosis.
* Anatomic obstructive voiding disorders
* Current urinary tract infection
* Malignancy of urinary tract
* Severe grade III/ IV pelvic prolapse, cystocele, urethrocele, enterocele
* Proven interstitial cystitis or clinical symptoms of interstitial cystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the eligibility for SNM therapy. This is defined as yes or no. A patient is eligible for the therapy when he or she can void again or the volume increased with at least 50%, and the catheterized volume is less then 100ml. | 3 weeks

SECONDARY OUTCOMES:
Complete or incomplete urinary retention | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip van Kerrebroeck, Professor, Principal Investigator — Maastricht University Hospital
Locations (1):
- dept Urology, Maastricht University Hospital, Maastricht, Netherlands